CLINICAL TRIAL: NCT00867672
Title: Prospective Randomized Multicenter Phase II Trial of Low-dose Decitabine (DAC) Administered Alone or in Combination With the Histone Deacetylase Inhibitor Valproic Acid (VPA) and All-trans Retinoic Acid (ATRA) in Patients > 60 Years With Acute Myeloid Leukemia Who Are Ineligible for Induction Chemotherapy
Brief Title: Study of Decitabine Alone or in Combination With Valproic Acid and All-trans Retinoic Acid in Acute Myeloid Leukemia
Acronym: DECIDER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Principal Investigator, Michael Luebbert, Professor, University Hospital Freiburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00332/AMLSG14-09
Record Dates: First submitted 2009-03-23; First posted 2009-03-24 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Low-dose Decitabine; Valproic acid; All-trans retinoic acid; Older Patients
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine; Valproic Acid; Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Decitabine (Experimental): i.v. Decitabine 20 mg/m² over 1h, 5 days (total dose 100 mg/m²), repeated every 4 weeks
  Interventions: Drug: Decitabine
- Decitabine+VPA (Experimental): i.v. Decitabine 20 mg/m² over 1h, 5 days (total dose 100 mg/m²), repeated every 4 weeks, and VPA (p.o.) from day 6 of first cycle continuously throughout all treatment cycles
  Interventions: Drug: Decitabine; Drug: VPA
- Decitabine+ATRA (Experimental): i.v. Decitabine 20 mg/m² over 1h, 5 days (total dose 100 mg/m²), repeated every 4 weeks and ATRA (45 mg/m² p.o.) from day 6 to day 28 of each treatment cycle
  Interventions: Drug: Decitabine; Drug: ATRA
- Decitabine+VPA+ATRA (Experimental): i.v. Decitabine 20 mg/m² over 1h, 5 days (total dose 100 mg/m²), repeated every 4 weeks and VPA (p.o.) from day 6 continuously throughout all treatment cycles and ATRA (45 mg/m² p.o.), from day 6 to day 28 of each treatment cycle
  Interventions: Drug: Decitabine; Drug: VPA; Drug: ATRA

INTERVENTIONS:
Drug: Decitabine — i.v. Decitabine 20 mg/m² over 1h, 5 days (total dose 100 mg/m²), repeated every 4 weeks
  Other Names: Dacogen
Drug: VPA — VPA starting on day 6 of first cycle continuously throughout all treatment cycles
  Other Names: Valproic acid
  Arms: Decitabine+VPA; Decitabine+VPA+ATRA
Drug: ATRA — ATRA (45 mg/m² p.o.) from day 6 to day 28 of each treatment cycle
  Other Names: All-trans retinoic acid
  Arms: Decitabine+ATRA; Decitabine+VPA+ATRA

SUMMARY:
AML of the older patient constitutes a major unmet clinical need since the large majority will not be found eligible for induction chemotherapy. Reasons for this decision include host factors (comorbidities, reduced performance status, functional limitations due to age), leading to often poor tolerance of repeated chemotherapy courses and the unfavorable biology underlying this disease in older patients. Low dose Decitabine has shown very promising efficacy in high-risk MDS and is therefore a very promising approach also in older AML patients. Preliminary results from several centres have demonstrated excellent feasibility and good efficacy of this treatment. Therefore the investigators intend to investigate the effects of two drugs added onto low-dose Decitabine which have shown very promising synergistic effects in vitro and for which preliminary results indicate that the combination with low-dose Decitabine is very feasible.

DETAILED DESCRIPTION:
By employing a 2x2 factorial design, this phase II study will address the possible added efficacy of addition of one or even both of these agents to low-dose Decitabine. The primary endpoint of this study will be objective response rate (complete and partial remissions).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained according to international guidelines and local law;
2. Male or female patients aged > 60 years without upper age limit;
3. Patients with primary or secondary AML according to WHO (≥ 20% blasts in the peripheral blood (pB) or bone marrow (BM)) who are not expected to benefit from standard remission-induction chemotherapy;
4. Patients with < 30 000 leukocytes/μl;
5. Performance status ECOG 0, 1, 2;
6. Creatinine < 2.0 mg/dl (unless leukemia-related);
7. Ability to understand the nature of the study and the study related procedures and to comply with them.

Exclusion Criteria:

1. AML of FAB subtype M3;
2. Previous remission-induction chemotherapy for MDS or AML, previous allografting;
3. Previous treatment with DAC, 5-azacytidine, VPA or another HDAC inhibitor, or ATRA;
4. "Low-dose" chemotherapy (e.g. hydroxyurea, cytosine arabinoside (Ara-C), melphalan, clofarabine etc.) within 4 weeks prior to DAC treatment, except for cytoreduction of leukocytosis ≥ 30 000/μl with hydroxyurea or Ara-C as proscribed by the study protocol (section 7.3 and 7.4); the patient must have recovered from all clinically relevant reversible non-hematologic toxicities;
5. Treatment with tyrosine kinase inhibitors, immunomodulating agents (IMIDS) or other investigational AML treatment within the last 4 weeks or in a time period of drug half-life x 5 (whatever is shorter) before the first administration of DAC;
6. Treatment with cytokines within previous 4 weeks;
7. Concomitant therapy which is considered relevant for the evaluation of efficacy or safety of the trial drug (i.e. other chemo- or immunotherapy);
8. Other malignancy requiring treatment (previous chemotherapy for other malignancies is not an exclusion criteria);
9. Cardiac insufficiency NYHA IV;
10. Insufficient hepatic function (bilirubin, AST or ALT > = 2.5 x Upper Limit of Normal (ULN)) (unless leukemia-related);
11. Fatal hepatic function disorder during treatment with valproic acid in siblings;
12. Hepatic porphyria;
13. Manifest serious pancreatic function disorder;
14. Plasmatic coagulation disorder not related to AML;
15. Known active hepatitis B or C;
16. Known HIV infection;
17. Other uncontrolled active infections;
18. Known allergy against soy beans or peanuts;
19. Psychiatric disorder that interferes with treatment;
20. Patient without legal capacity who is unable to understand the nature, significance and consequences of the study;
21. Known hypersensitivity to, or intolerance of, one of the trial drugs, another retinoid or the excipients of the trial drugs;
22. Concomitant use of any other investigational drug or participation in a clinical trial within the last thirty days before the start of this study; simultaneous participation in registry and diagnostic trials is allowed;
23. Female patients who are pregnant or breast feeding;
24. Fertile patients refusing to use safe contraceptive methods during the study (for details see clinical trial protocol section 5.3);
25. Known or persistent abuse of medication, drugs or alcohol.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2011-08; Primary Completion 2015-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Objective best response rate (complete remission (CR) and partial remission (PR)) | 12 months after randomization of the last patient

SECONDARY OUTCOMES:
Overall best response rate (CR, PR and antileukemic effect (ALE)) | 12 months after randomization of the last patient
progression-free survival (PFS) | 12 months after randomization of the last patient
overall survival (OS) | 12 months after randomization of the last patient
quality of life | until 4 weeks after study drug intake
safety and toxicity | until 4 weeks after study drug intake

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lübbert, MD, PhD, Principal Investigator — Department of Hematology/Oncology, University of Freiburg Medical Center
Locations (27):
- Germany (27):
  - Klinikum der Technischen Universität Aachen, Aachen
  - Vivantes Klinikum Neukölln, Berlin
  - Augusta-Kranken-Anstalt gGmbH, Bochum
  - Klinikum Braunschweig, Braunschweig
  - DIAKO Ev. Diakonie-Krankenhaus gGmbH, Bremen
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Marien Hospital Düsseldorf, Düsseldorf
  - Klinikum Esslingen GmbH, Esslingen am Neckar
  - Universität Frankfurt, Frankfurt
  - Medizinische Universitätsklinik Freiburg, Freiburg im Breisgau
  - St. Marien-Hospital Hagen, Hagen
  - Universitätsklinikum Halle, Halle
  - Evangelisches Krankenhaus Hamm gGmbH, Hamm
  - Med. Hochschule Hannover, Hanover
  - Universitätsklinikum Jena, Jena
  - Ortenau Klinikum Lahr-Ettenheim, Lahr
  - Caritas Krankenhaus Lebach, Lebach
  - Universitätsklinikum Leipzig AöR, Leipzig
  - Klinikum Lüdenscheid, Lüdenscheid
  - Philipps-Universität Marburg, Marburg
  - TU München, München
  - University of Münster Medical Center, Münster
  - Ortenau Klinikum, Offenburg
  - Studienzentrum Onkologie Ravensburg, Ravensburg
  - Eberhard Karls Universität Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - Klinikum Villingen-Schwenningen, Villingen-Schwenningen

REFERENCES:
- [Derived] Bresser H, Schmoor C, Grishina O, Pfeifer D, Thomas J, Rehman UU, Crysandt M, Jost E, Thol F, Heuser M, Gotze KS, Schlenk RF, Salih HR, Schittenhelm MM, Heil G, Schwaenen C, Muller-Tidow C, Brugger W, Kundgen A, de Wit M, Giagounidis A, Scholl S, Neubauer A, Krauter J, Bug G, May AM, Wasch R, Duyster J, Dohner K, Ganser A, Dohner H, Hackanson B, Becker H, Lubbert M. Impact of TP53 Mutation Status in Elderly AML Patients When Adding All-Trans Retinoic Acid or Valproic Acid to Decitabine. Eur J Haematol. 2025 Feb;114(2):231-237. doi: 10.1111/ejh.14304. Epub 2024 Oct 13. PMID 39400388
- [Derived] Thomas J, Rehman UU, Bresser H, Grishina O, Pfeifer D, Sollier E, Dohner K, Plass C, Becker H, Schmoor C, de Wit M, Lubbert M. Continued decitabine/all-trans retinoic acid treatment: extended complete remission in an elderly AML patient with multi-hit TP53 lesions and complex-monosomal karyotype. Clin Epigenetics. 2024 Sep 11;16(1):126. doi: 10.1186/s13148-024-01737-4. PMID 39261919
- [Derived] Javorniczky NR, Grishina O, Hund I, Pantic M, Pfeifer D, Schmoor C, Thomas J, Duyster J, Becker H, Lubbert M. Long-term decitabine/retinoic acid maintenance treatment in an elderly sAML patient with high-risk genetics. Clin Epigenetics. 2023 Nov 28;15(1):185. doi: 10.1186/s13148-023-01596-5. PMID 38012682
- [Derived] Lubbert M, Grishina O, Schmoor C, Schlenk RF, Jost E, Crysandt M, Heuser M, Thol F, Salih HR, Schittenhelm MM, Germing U, Kuendgen A, Gotze KS, Lindemann HW, Muller-Tidow C, Heil G, Scholl S, Bug G, Schwaenen C, Giagounidis A, Neubauer A, Krauter J, Brugger W, De Wit M, Wasch R, Becker H, May AM, Duyster J, Dohner K, Ganser A, Hackanson B, Dohner H; DECIDER Study Team. Valproate and Retinoic Acid in Combination With Decitabine in Elderly Nonfit Patients With Acute Myeloid Leukemia: Results of a Multicenter, Randomized, 2 x 2, Phase II Trial. J Clin Oncol. 2020 Jan 20;38(3):257-270. doi: 10.1200/JCO.19.01053. Epub 2019 Dec 3. PMID 31794324
- [Derived] Grishina O, Schmoor C, Dohner K, Hackanson B, Lubrich B, May AM, Cieslik C, Muller MJ, Lubbert M. DECIDER: prospective randomized multicenter phase II trial of low-dose decitabine (DAC) administered alone or in combination with the histone deacetylase inhibitor valproic acid (VPA) and all-trans retinoic acid (ATRA) in patients >60 years with acute myeloid leukemia who are ineligible for induction chemotherapy. BMC Cancer. 2015 May 26;15:430. doi: 10.1186/s12885-015-1432-5. PMID 26008690
- See also: Study protocol publication — https://bmccancer.biomedcentral.com/articles/10.1186/s12885-015-1432-5